CLINICAL TRIAL: NCT00270478
Title: Evaluation of Synergy of Combining Hydroxyurea With Recombinant Human Erythropoietin Glycoform Alpha (Rhu Erythropoietin-alpha) on Fetal Hemoglobin Synthesis in Patients With Sickle Cell Anemia
Brief Title: Hydroxyurea and Erythropoietin to Treat Sickle Cell Anemia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 060054; 06-H-0054
Record Dates: First submitted 2005-12-25; First posted 2005-12-26 (Estimated); Last update posted 2019-12-17 (Actual); Status verified 2016-01-27

CONDITIONS: Sickle Cell Disease; Chronic Kidney Disease; Pulmonary Hypertension
Keywords: Erythropoietin Therapy; Fetal Hemoglobin Induction; Sickle Cell Disease; Pulmonary Hypertension; Chronic Kidney Disease; SCD
MeSH Terms: conditions — Anemia, Sickle Cell; Renal Insufficiency, Chronic; Hypertension, Pulmonary | interventions — Erythropoietin; Hydroxyurea

INTERVENTIONS:
Drug: Erythropoietin and Hydroxyurea

SUMMARY:
This study will examine the use of hydroxyurea and erythropoietin for treating sickle cell disease in patients who also have kidney disease or pulmonary hypertension (high blood pressure in the lungs). Hydroxyurea increases production of fetal hemoglobin in the red blood cells of patients with sickle cell disease, reducing the amount of sickle cells that cause pain and other complications requiring hospitalizations. However, hydroxyurea treatment has limitations: patients with sickle cell disease who have developed kidney disease may not be able to get the full benefit of the medicine, and hydroxyurea alone may not be able to treat life-threatening complications such as pulmonary hypertension or stroke. This study will determine which of two dosing schedules of hydroxyurea and erythropoietin is more effective for treating patients with sickle cell disease who also have kidney disease or pulmonary hypertension, and will examine whether the two drugs can lower blood pressure in the lungs.

Patients 18 years of age and older with sickle cell anemia and kidney disease or pulmonary hypertension, or both, may be eligible for this study. Candidates are screened with a medical history, physical examination, blood tests, a 6-minute walk test (test to see how far the subject can walk in 6 minutes), and echocardiogram (ultrasound of the heart to measure blood pressure in the lungs).

Participants undergo the following tests and procedures:

Stabilization Phase: Patients take 2 hydroxyurea tablets a day until their fetal hemoglobin levels stabilize, usually over 2 to 4 months. They have blood tests every 2 weeks to monitor hemoglobin and fetal hemoglobin levels. At some time during this period, they undergo a test to measure kidney function, in which they are injected with an iodine-containing dye and wear a small pump for 1 day that injects a small amount of dye under the skin over 24 hours. They come to the clinic for 2 or 3 blood tests collected over 4 hours.

Sequence I (Standard): When the fetal hemoglobin levels have been stable for 2 months, patients have a repeat echocardiogram and 6-minute walk test. Erythropoietin is then added to the hydroxyurea regimen. It is given 3 days a week, as an injection under the skin, along with iron supplements. Patients have blood tests and blood pressure measurements every week or every other week. Patients with pulmonary hypertension have another echocardiogram and 6-minute walk test once the hemoglobin level is stable.

Sequence II (Cycled): When hemoglobin levels have stabilized with hydroxyurea once a day and erythropoietin 3 times a week, the hydroxyurea is adjusted so that the amount taken in 7 days is "cycled" over 4 days, and the erythropoietin is cycled over 3 days, with the dose increased twice, every 3 to 4 weeks. Blood pressure and hemoglobin are monitored once or twice a month. Patients with pulmonary hypertension have another echocardiogram and 6-minute walk test once the hemoglobin level is stable.

Patients who develop complications while taking the drugs have their treatment regimens adjusted as needed.

DETAILED DESCRIPTION:
Sickle cell disease (SCD) is a genetic disease that afflicts over eighty thousand Americans, 4 to 5,000 newborns per year in the US, and 100s of thousands of children and adults world-wide. This disease arises from a single amino acid mutation of the beta globin chain of hemoglobin, which results in abnormal polymerization of deoxygenated hemoglobin. The deceptively simple biologic origin for SCD belies the debilitating chronic multi-faceted clinical syndrome with which it is associated; SCD is characterized by lifelong hemolysis, chronic anemia, recurrent painful vaso-occlusive crises (VOC), hepatic, renal, musculo-skeletal, and central nervous system complications, and a shortened life-expectancy. Our group has found an up to 33% incidence of pulmonary hypertension in adult patients with SCD who were screened and followed prospectively; with two-year follow-up, this pulmonary hypertension is associated with a 10-fold increased mortality rate.

Hydroxyurea has emerged as a useful therapy in sickle cell disease. It is a cell-cycle specific agent that blocks DNA synthesis by inhibiting ribonucleotide reductase, the enzyme that converts ribonucleotides to deoxyribonucleotides. Hydroxyurea has been shown to induce the production of fetal hemoglobin (HbF) in patients with sickle cell anemia, with associated diminished morbidity and, likely, mortality in these patients. Any HbF is good in SCD, although it is estimated that levels of 20 percent HbF are required to substantially reduce the sickling propensity of red cells and to modulate disease severity. The majority of patients with SCD respond to hydroxyurea with a more than two-fold increase in HbF levels; in some patients the percent of HbF exceeds 10 or 15 percent, but it is not uniformly distributed in all cells, i.e. has a hetero-cellular rather than a pan-cellular distribution. The mechanism through which hydroxyurea augments fetal Hgb is incompletely characterized. An additional benefit of hydroxyurea may be through effects on the nitric oxide (NO) system. Recently, members of our group found that hydroxyurea therapy is associated with the intravascular and intra-erythrocytic generation of NO, and that NO increases HbF expression via the guanylyl cyclase/cGMP dependent pathways.

We have treated more than 30 patients chronically with hydroxyurea to determine hematological changes Iongitudinally, and have established the maximal HbF raising effect of hydroxyurea in these patients. We have found that the levels of HbF that are induced by hydroxyurea alone are insufficient, and insufficiently widely distributed, to ameliorate the life-threatening complications of pulmonary HTN and of on-going hemolysis in patients with sickle cell disease.

Earlier studies had suggested that the addition of erythropoietin (Erythropoietin) therapy to chronic hydroxyurea therapy may induce fetal hemoglobin at higher, more widely distributed, levels. We plan to test this in patients with sickle cell disease who have chronic kidney disease, which, presumably, leaves them with a depressed Erythropoietin reserve and an inability to tolerate standard doses of F-inducing therapy with hydroxyurea, and in patients with pulmonary HTN, which carries an ominous prognosis in SCD. A secondary endpoint of this study will be to evaluate if hydroxyurea plus Erythropoietin therapy can improve cardiovascular aerobic capacity in general, and in particular minimize symptoms and morbidity in patients with both chronic kidney disease and pulmonary HTN.

ELIGIBILITY:
* INCLUSION CRITERIA:

Patients with homozygous SCD or other sickling disorders (e.g., B(0) Thalassemia/Sickle) who are 18 years of age or greater will be eligible for treatment. Patients currently being followed on an NIH study or at Howard University on stable doses of hydroxyurea are also eligible. A total of 60 patients will be recruited to the study, with the recognition from our earlier studies of a failure-to-complete rate approaching 50%.

Patients must have documented hemoglobin S-only or S-beta(0)-thalassemia.

Patients must have relatively well preserved hepatic function (less than 3 X upper limits of normal ALT).

Patients must be able to provide informed consent.

Patients must have:

-an eGFR of 15 to 60 ml/min per 1.73 m(2) BSA,

or

an eGFR of 61 - 90 ml/min per 1.73 m(2) BSA and greater than 16.9 mg of albumin/g creatinine (greater than 0.017 ratio g/g),

and/or

a trans-thoracic echocardiographic measurements of pulmonary artery pressure (PAP), as estimated by tricuspid regurgitant velocity, of greater than 2.5 m sec(-1) monthly at baseline times two.

EXCLUSION CRITERIA:

Patients who are doubly heterozygous for hemoglobin-S and fully or partially expressed hemoglobin-A or any other non-S beta-type globin chain, or hemoglobin A-only (non-sickle cell).

Patients who are on a chronic transfusion program, defined as regular transfusions every 2-8 weeks.

Patients who are pregnant or breast-feeding.

Patients who have a history of a documented cerebrovascular accident or venous thrombosis within one year of study entry.

Patients with active proliferative retinopathy within 1 year of study entry

Patients with eGFR less than or equal to 14 ml/min per 1.73 M(2) BSA.

Patients with a total Hgb at entry that is 10.5 g/dl or greater

Patients with a known allergy to Albumin or cell-derived products

Patients with uncontrolled hypertension, defined as a systolic blood pressure greater than 170 mmHg and diastolic blood pressure greater than 110 mm Hg that is sustained and unresponsive over 1 week to conventional anti-hypertensive therapy .

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2005-12-21; Primary Completion 2009-08-31 (Actual); Study Completion 2009-08-31 (Actual)

PRIMARY OUTCOMES:
An increase in fetal hemoglobin, as measured by high performance liquid chromatograph, from hydroxyurea alone/stabilized baseline to concurrent Erythropoietin in standard therapy/sequence l.

SECONDARY OUTCOMES:
(All measured, at a minimum, at study entry, at change of dose, and with stabilization at the conclusion of each Erythropoietin sequence, standard or cycled).

CONTACTS AND LOCATIONS:
Overall Officials: John F Tisdale, M.D., Principal Investigator — National Heart, Lung, and Blood Institute (NHLBI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Platt OS, Thorington BD, Brambilla DJ, Milner PF, Rosse WF, Vichinsky E, Kinney TR. Pain in sickle cell disease. Rates and risk factors. N Engl J Med. 1991 Jul 4;325(1):11-6. doi: 10.1056/NEJM199107043250103. PMID 1710777
- [Background] Platt OS, Brambilla DJ, Rosse WF, Milner PF, Castro O, Steinberg MH, Klug PP. Mortality in sickle cell disease. Life expectancy and risk factors for early death. N Engl J Med. 1994 Jun 9;330(23):1639-44. doi: 10.1056/NEJM199406093302303. PMID 7993409
- [Background] McKerrell TD, Cohen HW, Billett HH. The older sickle cell patient. Am J Hematol. 2004 Jun;76(2):101-6. doi: 10.1002/ajh.20075. PMID 15164373